CLINICAL TRIAL: NCT05540600
Title: Left Atrium Reservoir Function Modulation in Patients With Atrial Fibrillation: A Randomized Digoxin Versus Beta Blocker Study
Brief Title: Left Atrium Reservoir Function Modulation in Patients With Atrial Fibrillation: Digoxin Versus Beta Blocker
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Nidhal Bouchahda, Principal investigator, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TN2022-NAT-I NS-86
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation; Left Atrial Rhythm
MeSH Terms: conditions — Atrial Fibrillation | interventions — Digoxin; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digoxin group (Experimental): Patients will receive digoxin 0.25 mg once daily for a duration of 4 weeks
  Interventions: Drug: Digoxin 0.25 mg
- beta blocker group (Experimental): Patients will receive bisoprolol 2.5 mg or 5 m twice a day for a duration of 4 weeks. The choice of dose will depend on blood pressure (BP): If systolic BP ≥ 150 mmHG, the patient will have bisoprolol 5 mg x 2 per day, If systolic BP < 150 mmHG, the patient will have bisoprolol 2.5 mg x 2 per day
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Digoxin 0.25 mg — Patients will have the dose of one tablet of 0.25mg per day
  Arms: Digoxin group
Drug: Bisoprolol — Patients will have the dose of bisoprolol 2.5 mg or 5 mg twice a day based on the arterial pressure at randomization
  Arms: beta blocker group

SUMMARY:
ß blocker and digoxin effect on left atrium reservoir function are unknown. This is a randomized open label study to compare the effect of theses two molecules on left atrium function

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is responsible of significant morbidity and mortality. Management of signs and symptoms of heart failure generated by AF is at the center of the latest European recommendations . Mechanisms by which these symptoms are generated are very poorly understood. Heart rate control is one of the recommended strategies but remains poorly codified and generally follows the preferences and experiences of each local center. The European guidelines propose at least 4 molecules for heart rate control without emitting preferences for one molecule over the other due to the lack of robust randomized studies. Recently, a study comparing digoxin vs ß-blockers showed the superiority of digoxin in decreasing symptoms despite a comparable action on heart rate. On the other hand, the reservoir function of the left atrium (LA) has taken a central role in assessing signs of left heart failure and monitoring filling pressures . Other studies have demonstrated the association of left atrium reservoir strain with these symptoms .

It is commonly accepted that ß blockers decrease AF-related symptoms by a negative chronotropic effect thanks to their blocking action on the sympathetic system. While the action of digoxin on symptoms goes through a positive inotropic effect thanks to the increase in intracellular calcium .

However, the impact of these two molecules on the function of the left atrium has never been investigated. Our diagnostic hypothesis is that in addition to their action on heart rate, the improvement of symptoms noted by using b blockers and digoxin during the treatment of AF would go through an improvement LA reservoir function . The superiority of digoxin in the reduction of symptoms compared to ß blockers would be due to a greater improvement in reservoir function and this thanks to the increase in myocardial intracellular calcium.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with atrial fibrillation naïve to ß-blocker and digoxin or patients followed for Atrial fibrillation and discontinued all treatment for more than a week.
* Frequency Control Strategy Decided
* Age over 18 years
* Stable hemodynamic state
* No contraindication to digoxin or ß-blocker

Exclusion Criteria:

* Required rhythm control strategy
* Contraindication to one of the two
* Heart rate <60 BPM
* Clearance rénale <30 ml/mn
* Pregnant or breastfeeding woman
* Persistence of a resting heart rate > 110
* Severe comorbidity with decreased life expectancy (advanced neoplasia, large stroke...)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Left atrium reservoir strain before and after treatment | 4 weeks
  Measurements of Left atrium reservoir strain will be performed at randomization and after 4 weeks on 4 chambers and 2 chamber views according to the most recent recommendations. The acquisition of strain-2D curves will be made by taking as a reference the beginning of the QRS complex. The peak of the curve corresponds to the value of the reservoir strain of the left atrium

CONTACTS AND LOCATIONS:
Overall Officials: Nidhal Bouchahda, MD, Principal Investigator — Monastir university
Locations (1):
- Fattouma Bourguiba University hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotecha D, Bunting KV, Gill SK, Mehta S, Stanbury M, Jones JC, Haynes S, Calvert MJ, Deeks JJ, Steeds RP, Strauss VY, Rahimi K, Camm AJ, Griffith M, Lip GYH, Townend JN, Kirchhof P; Rate Control Therapy Evaluation in Permanent Atrial Fibrillation (RATE-AF) Team. Effect of Digoxin vs Bisoprolol for Heart Rate Control in Atrial Fibrillation on Patient-Reported Quality of Life: The RATE-AF Randomized Clinical Trial. JAMA. 2020 Dec 22;324(24):2497-2508. doi: 10.1001/jama.2020.23138. PMID 33351042
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P, Agewall S, Camm J, Baron Esquivias G, Budts W, Carerj S, Casselman F, Coca A, De Caterina R, Deftereos S, Dobrev D, Ferro JM, Filippatos G, Fitzsimons D, Gorenek B, Guenoun M, Hohnloser SH, Kolh P, Lip GY, Manolis A, McMurray J, Ponikowski P, Rosenhek R, Ruschitzka F, Savelieva I, Sharma S, Suwalski P, Tamargo JL, Taylor CJ, Van Gelder IC, Voors AA, Windecker S, Zamorano JL, Zeppenfeld K. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur J Cardiothorac Surg. 2016 Nov;50(5):e1-e88. doi: 10.1093/ejcts/ezw313. Epub 2016 Sep 23. No abstract available. PMID 27663299
- [Background] Ziff OJ, Kotecha D. Digoxin: The good and the bad. Trends Cardiovasc Med. 2016 Oct;26(7):585-95. doi: 10.1016/j.tcm.2016.03.011. Epub 2016 Mar 31. PMID 27156593
- [Background] Badano LP, Kolias TJ, Muraru D, Abraham TP, Aurigemma G, Edvardsen T, D'Hooge J, Donal E, Fraser AG, Marwick T, Mertens L, Popescu BA, Sengupta PP, Lancellotti P, Thomas JD, Voigt JU; Industry representatives; Reviewers: This document was reviewed by members of the 2016-2018 EACVI Scientific Documents Committee. Standardization of left atrial, right ventricular, and right atrial deformation imaging using two-dimensional speckle tracking echocardiography: a consensus document of the EACVI/ASE/Industry Task Force to standardize deformation imaging. Eur Heart J Cardiovasc Imaging. 2018 Jun 1;19(6):591-600. doi: 10.1093/ehjci/jey042. PMID 29596561
- [Derived] Bouchahda N, Bader M, Najjar A, Mghaieth Zghal F, Sassi G, Mourali MS, Ben Messaoud M. Effect of Digoxin vs Beta-Blockers on Left Atrial Strain for Heart Rate-Controlled Atrial Fibrillation: The DIGOBET-AF Randomized Clinical Trial. Am J Cardiovasc Drugs. 2025 May;25(3):411-418. doi: 10.1007/s40256-024-00705-w. Epub 2024 Dec 26. PMID 39725795